CLINICAL TRIAL: NCT00005604
Title: Phase I Trial of Twice Weekly IV IL-12 Plus Low-Dose Subcutaneous IL-2 in Patients With Advanced Malignancies
Brief Title: Interleukin-12 Plus Interleukin-2 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00049; BIDMC #99-1332; CDR0000067723 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-05-02; First posted 2003-07-24 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Interleukin-12 Subunit p35; Interleukin-12; aldesleukin; Interleukin-2

ARMS (1):
- Treatment (rhIl-12, IL-2) (Experimental): Patients receive interleukin-12 (IL-12) IV on days 1 and 4 for 6 weeks. Beginning on day 4 of the third week, patients receive interleukin-2 (IL-2) subcutaneously 1 hour before and 20 hours after each dose of IL-12. On subsequent courses, IL-2 and IL-12 are administered on days 1 and 4 of each week. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease response may continue treatment until complete response or disease progression.
  Interventions: Biological: recombinant interleukin-12; Biological: aldesleukin; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant interleukin-12 — Given IV
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of interleukin-12 plus interleukin-2 in treating patients who have advanced solid tumors. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining the two drugs may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity profile and MTD of low-dose SC IL-2 administered in conjunction with BIW regimen of IV rhIL-12.

II. To determine the antitumor effects of combination therapy with IV rhIL-12 and SC IL-2.

III. To determine the impact low-dose SC IL-2 has on the magnitude and duration of in vivo immune activation induced by a BIW schedule of IV rhIL-12.

OUTLINE: This is a dose-escalation study.

Patients receive interleukin-12 (IL-12) IV on days 1 and 4 for 6 weeks. Beginning on day 4 of the third week, patients receive interleukin-2 (IL-2) subcutaneously 1 hour before and 20 hours after each dose of IL-12. On subsequent courses, IL-2 and IL-12 are administered on days 1 and 4 of each week. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease response may continue treatment until complete response or disease progression.

Cohorts of 3-6 patients receive escalating doses of IL-12 and IL-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed solid tumor malignancy which is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; patients with hematologic malignancies will be excluded
* Patients must have advanced measurable or evaluable disease which is clearly progressive
* Patients must be ambulatory with good performance status (ECOG PS 0 or 1; Karnofsky PS 100-80%) and have an anticipated survival of at least 3 months
* Women of child bearing potential must have a negative pregnancy test and will be expected to use proven contraceptive methods while on protocol therapy; women who are breast-feeding are excluded from this study
* WBC > 4000/mm^3
* ANC > 1500/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 1.5 mg/dl
* SGOT, SGPT < 2 x normal
* Creatinine < 1.5 mg/dl or calculated creatinine clearance >= 60 ml/min
* No evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmias, or evidence of prior myocardial infarction on EKG
* No evidence of active infection which requires antibiotic therapy or history of treatment with IV antibiotics for a documented infection within 2 weeks of beginning treatment
* Patients must have recovered from the toxicity of prior therapy and have clearly progressive disease
* CHEMO, HORMONAL, AND RADIOTHERAPY There is a limit of two prior chemotherapy regimens which patients may have received; (patients who have received extensive prior cytotoxic therapy may no longer have adequate organ function and may not be eligible); at least 4 weeks must have elapsed from the end of previous chemotherapy, hormonal therapy, or radiotherapy (six weeks for nitrosoureas or mitomycin); concurrent chemotherapy, hormonal therapy or radiotherapy is not permitted; patients on steroids, including replacement therapy, will be excluded from the study
* BIOLOGICAL RESPONSE MODIFIERS No more than 2 prior BRM treatment regimens are permitted; prior immunotherapy should have been completed at least 4 weeks prior to beginning treatment on this protocol; prior therapy will IL-2 or rhIL-12 is allowable if >= 6 months have elapsed since the end of IL-2 treatment or if >= 12 months have elapsed since rhIL-12 therapy
* The patient must give signed informed consent prior to the initiation of therapy; patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with therapy
* Patients with the following problems will be considered ineligible:

  * Organ allografts

    * Brain metastases
    * Seizure disorders
    * Patients known to be HIV positive are excluded based on the potential harm these agents may have on their underling immune function and the unknown effects of combination therapy with IL-12 and IL-2 on HIV viral replication; in addition, HIV infection, through its documented deleterious effects on lymphocyte number and function, may impair the patient's ability to respond to this form of cytokine-based immunotherapy
    * Any medical condition likely to require use of corticosteroids during IL-12 therapy
    * Autoimmune or rheumatologic disease
    * Active (clinical or subclinical) hepatitis B or hepatitis C infection
    * Any significant medical disease other than the malignancy felt by the investigator to place the patient at greater risk for developing a life-threatening toxicity from the therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-03; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level that is just below the dose on which at least 2 of 6 patients developed a dose-limiting toxicity (DLT) as assessed by CTC version 2.0 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Atkins, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States